CLINICAL TRIAL: NCT00982683
Title: Association of Lunar Phases With Post-surgical Hemorrhagic Rate
Brief Title: Association of Lunar Phases With Post-surgical Morbidity
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: University of Genova (Other)
Responsible Party: Edoardo Raposio, MD, PhD, FICS, National Institute for Cancer Research, Genova, Italy
Other Study IDs: Moon-01
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Hemorrhage
Keywords: Surgery; Moon phases; hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The potential influence of lunar phases on human life has been widely discussed by the lay press. The purpose of this study was to evaluate a possible relation between the lunar cycle and the hemorrhagic complication rate and surgical outcome.

PATIENTS AND METHODS:

The investigators tested this hypothesis by evaluating the complication rate for 18760 patients who underwent surgery from January 2001 to December 2008 (103 lunar phases) at the National Institute for Cancer Research in Genoa.

The date of definitive surgery was allocated to the lunar phases.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated at the National Cancer Institute, Genoa, Italy, during the period 2001-2008
Sampling Method: Non-Probability Sample
Enrollment: 26244 (Actual)
Dates: Start 1998-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Dependence analysis between post-surgical complications and lunar phases. | 2001 - 2008

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Raposio, MD, Principal Investigator — National Cancer Institute, Italy
Locations (1):
- National Cancer Institute, Italy, Genova, Italy

REFERENCES:
- [Background] Sha LR, Xu NT, Song XH, Zhang LP, Zhang Y. Lunar phases, myocardial infarction and hemorrheological character. A Western medical study combined with appraisal of the related traditional Chinese medical theory. Chin Med J (Engl). 1989 Sep;102(9):722-5. PMID 2517088